CLINICAL TRIAL: NCT02725346
Title: ArthroPlanner: A Surgical Planning Solution for Acromioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, MD, La Tour Hospital
Organization: La Tour Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GE 15-151
Record Dates: First submitted 2016-03-11; First posted 2016-04-01 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Shoulder Impingement Syndrome; Subacromial Impingement Syndrome; Tendon Injuries
Keywords: Surgical Planning Solution; Acromioplasty; Shoulder Surgery; Critical Shoulder Angle
MeSH Terms: conditions — Shoulder Impingement Syndrome; Tendon Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-assisted planning (Experimental): Acromioplasty with planification
  Interventions: Procedure: Acromioplasty with planning
- No planning (Active Comparator): Acromioplasty without planification
  Interventions: Procedure: Acromioplasty without planning

INTERVENTIONS:
Procedure: Acromioplasty with planning
  Arms: Computer-assisted planning
Procedure: Acromioplasty without planning
  Arms: No planning

SUMMARY:
A computer-assisted solution for acromioplasty is presented. The software allows surgeons to better plan the surgical procedure by visualizing dynamic simulation of the patient's shoulder joint during everyday activities. Impingements are dynamically detected and the exact location and amount of bone to be resected is precisely computed. As a result, the success of the acromioplasty does not only rely on the surgeon's experience or previous recommendations, but on quantitative data. Although the clinical validation of this 3D planning support is currently under evaluation, it may allow to recover more effectively postoperative joint mobility, to get a better relationship with pain and a better healing rate of the rotator cuff tendons.

DETAILED DESCRIPTION:
Introduction Subacromial impingement of the rotator cuff between the anterior [1] or lateral acromion [2] and the superior humeral head is a common disorder. This condition arises when the subacromial space height is too narrow during active elevation or scaption of the arm above shoulder level due to an abnormal hooked shape or large lateral extension of the acromion.

In severe cases of impingement syndrome, an arthroscopic acromioplasty surgery is usually performed to resect the different area of the acromion causing damage to the subacromial structures. The exact location and the amount of bone to be resected is generally left to the unique appreciation of the orthopedic surgeon during surgery. To improve the precision of this resection, surgeons could greatly benefit from a surgical planning solution that aims at providing precise information about the surgical procedure. Moreover, since subacromial impingements are the result of a dynamic mechanism, an effective planning solution should analyze both the morphological joint's structures and its dynamic behavior during shoulder movements to fully apprehend the patient joint's condition.

Computer-assisted planning solution "ArthroPlanner" for acromioplasty is nowadays available. The solution allows to perform standard morphological bony measurements, as well as 3D simulations of the patient's joint during everyday shoulder activities. The software computes the precise bone resection (location and amount) based on detected subacromial impingements during motion.

The goal of this study was thus to compare clinical and radiological results of superior rotator cuff repair with or without computer-assisted planning. The hypothesis was that preoperative planning of acromioplasty would allowed more accurate bone resection, would decrease postoperative impingements and consequently improved postoperative range of motion and tendon healing.

Methods

We reconstruct the bones of the patient's shoulder joint (scapula and humerus from the humeral head to the mid-shaft) from a CT image using Mimics software (Materialise NV, Leuven, Belgium). The bones are then imported into ArthroPlanner software and the following steps are performed:

First, generic bone models are produced using a template fitting approach that deforms a bone template with an optimized topology (one for the scapula and one for humerus) to the reconstructed bone. This allows us in the next steps to exploit anatomical correspondences and to automatize landmarks and points selection on the mesh.

Second, biomechanical parameters are computed to permit motion description of the glenohumeral joint. The glenohumeral joint center is automatically calculated by a sphere fitting technique [3] that fits a sphere to the humeral head using the points of the proximal humerus model. Bone coordinate systems are established for the scapula and humerus. based on the definitions suggested by the International Society of Biomechanics [4] using anatomical landmarks defined on the bone models. Missing landmarks such as the lateral and medial epicondyles are identified on the CT image.

Third, morphological measurements are performed to analyze individual shoulder anatomy. The Critical Shoulder Angle [5] and the β angle [6] are calculated, as they are criteria associated with rotator cuff tears. The angles are computed in 3D based on bony landmarks and can be, if necessary, interactively adjusted by the user by manipulating 3D handles in the viewer.

Fourth, motion is applied at each time step to the humerus model with real-time evaluation of impingement. The minimum humero-acromial distance that is typically used for the evaluation of subacromial impingement is measured [7]. This distance is calculated in millimeters based on the simulated bones models positions. A color scale is also used to map the variations of distance on the scapula surface (red color = minimum distance, other colors = areas of increased distance). Given the thickness of the potential impinged tissues, subacromial impingement is considered when the computed humero-acromial distance is < 6 mm, as suggested in the literature [7]. To test a wide variability of realistic movements, a motion database of daily activities (e.g., cross arm, comb hair) is used in addition to standard kinematic sequences (e.g., elevation, scaption).

Finally, the acromial resection plan is defined based on the 3D simulation results. A color map is used to represent areas where impingements occurred between the acromion and humerus (Fig. 1D). The red color denotes the area with the smallest humero-acromial distance computed over the different motion simulations.

The results at each step of the planning procedure are carefully validated by the user before continuing to the next ones. At the end of the planning, a PDF report is generated that contains patient's information and the measurements performed. The bones and the simulation data are also exported to be used in a simple 3D viewer (Fig. 2) dedicated to the surgeon. With this viewer, the surgeon is able to play all simulations, observe impingements dynamically and review the resection plan.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic supraspinatus repair

Exclusion Criteria:

* Incomplete documentation
* Follow-up of less than six months
* Previous shoulder surgery
* Contraindications for computed tomography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Volume in mm3 of bone removal in four zones determine between pre- and postoperative computed tomography | 6 months
  Accuracy of acromioplasty in relation to preoperative planning (zone 1 anterior, zone 2 lateral, zone 3 medial, zone 4 central).
Tendon healing determine with ultrasound with Sugaya criteria | 6 month
  ultrasound realized by a blinded radiologist. This outcome will be considered as primary only if the first primary outcome is reached. Otherwise it will considered as a secondary outcome.

SECONDARY OUTCOMES:
Percentage of gain of range of motion between groups of postoperative range of motion | 6 month
  Evaluated by a independent and blind observer with dedicated software
Constant score | 6 months
American Shoulder and Elbow Surgeons score | 6 months
Simple shoulder value | 6 months
Single Assessment Numeric Evaluation score | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450
- [Background] Nyffeler RW, Werner CM, Sukthankar A, Schmid MR, Gerber C. Association of a large lateral extension of the acromion with rotator cuff tears. J Bone Joint Surg Am. 2006 Apr;88(4):800-5. doi: 10.2106/JBJS.D.03042. PMID 16595470
- [Background] Wu G, van der Helm FC, Veeger HE, Makhsous M, Van Roy P, Anglin C, Nagels J, Karduna AR, McQuade K, Wang X, Werner FW, Buchholz B; International Society of Biomechanics. ISB recommendation on definitions of joint coordinate systems of various joints for the reporting of human joint motion--Part II: shoulder, elbow, wrist and hand. J Biomech. 2005 May;38(5):981-992. doi: 10.1016/j.jbiomech.2004.05.042. PMID 15844264
- [Background] Moor BK, Bouaicha S, Rothenfluh DA, Sukthankar A, Gerber C. Is there an association between the individual anatomy of the scapula and the development of rotator cuff tears or osteoarthritis of the glenohumeral joint?: A radiological study of the critical shoulder angle. Bone Joint J. 2013 Jul;95-B(7):935-41. doi: 10.1302/0301-620X.95B7.31028. PMID 23814246
- [Background] Daggett M, Werner B, Collin P, Gauci MO, Chaoui J, Walch G. Correlation between glenoid inclination and critical shoulder angle: a radiographic and computed tomography study. J Shoulder Elbow Surg. 2015 Dec;24(12):1948-53. doi: 10.1016/j.jse.2015.07.013. Epub 2015 Sep 6. PMID 26350880
- [Background] Charbonnier C, Chague S, Kolo FC, Ladermann A. Shoulder motion during tennis serve: dynamic and radiological evaluation based on motion capture and magnetic resonance imaging. Int J Comput Assist Radiol Surg. 2015 Aug;10(8):1289-97. doi: 10.1007/s11548-014-1135-4. Epub 2014 Dec 14. PMID 25503926